CLINICAL TRIAL: NCT04820829
Title: Effects of Proportioning Meat and Plant-based Protein-rich Foods Within the U.S. Healthy Eating Pattern on Cardiovascular Disease Risk Factors (S58)
Brief Title: Effects of Proportioning Meat and Plant-based Protein-rich Foods on Cardiovascular Disease Risk Factors (S58)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: IRB-2020-587
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Healthy Diet; Cardiovascular Risk Factor
Keywords: Healthy eating pattern

STUDY DESIGN:
Intervention Model Description: The Investigator will use a randomized, cross-over (balanced incomplete block) experimental design, with separate randomizations for males and females. All participants will consume a U.S. HEP - all foods provided - during 5-week controlled feeding periods. Each participant will complete two of the three controlled feeding periods, separated by four weeks when they will consume their usual unrestricted diet (washout). The three HEP interventions will be: high RM, low NSS; moderate RM, moderate NSS; and low RM, high NSS. Measurements will be made before (usual unrestricted diet) and during the last week of each HEP intervention.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High RM, low NSS (Active Comparator): Participants in this group will consume nine 3-oz-eq servings of RM per week and 2-oz-eq servings of NSS per week.
  Interventions: Other: High RM, low NSS
- Moderate RM, moderate NSS (Active Comparator): Participants in this group will consume five 3-oz-eq servings of RM per week and 5-oz-eq servings of NSS per week.
  Interventions: Other: Moderate RM, Moderate NSS
- Low RM, high NSS (Active Comparator): Participants in this group will consume one 3-oz-eq serving of RM per week and 8-oz-eq servings of NSS per week.
  Interventions: Other: Low RM, High NSS

INTERVENTIONS:
Other: High RM, low NSS — Participants in this group will consume nine 3-oz-eq servings of RM per week and 2-oz-eq servings of NSS per week.
  Arms: High RM, low NSS
Other: Moderate RM, Moderate NSS — Participants in this group will consume five 3-oz-eq servings of RM per week and 5-oz-eq servings of NSS per week.
  Arms: Moderate RM, moderate NSS
Other: Low RM, High NSS — Participants in this group will consume one 3-oz-eq serving of RM per week and 8-oz-eq servings of NSS per week.
  Arms: Low RM, high NSS

SUMMARY:
This project will assess the effects of consuming different proportions of red meat (RM) and plant-based, protein-rich foods (nuts, seeds, and soy products - NSS) incorporated into a U.S. Healthy Eating Pattern (HEP) on cardiovascular disease risk factors in adults at high risk of developing a heart-related disease.

DETAILED DESCRIPTION:
Using a randomized, cross-over (balanced incomplete block) experimental design, Forty-eight middle-aged adults who are overweight and have high blood total cholesterol and LDL-C concentrations will be recruited. Participants will consume a HEP - all foods provided - during 5-week controlled feeding periods. The three HEP interventions will be: high RM, low NSS; moderate RM, moderate NSS; and low RM, high NSS. Each participant will complete two of the three controlled feeding periods, separated by four weeks when participants will consume their usual unrestricted diet (washout). The HEP consumed during the controlled feeding periods will be the same except for the amounts of RM (1, 5, or 9, 3-oz servings/wk) and NSS (high, moderate, and low, with amounts adjusted to isocalorically offset changes in RM energy intakes). Poultry, egg, and legume intakes will be the same among the three HEP. The investigators will measure clinically important cardiovascular disease risk factors before (usual unrestricted diet) and during the last week of each HEP intervention. The cardiovascular disease risk factors will include, but are not limited to, comprehensive lipid and lipoprotein profile (changes in low-density lipoprotein cholesterol, LDL-C; primary outcome), lipoprotein fractionation and particle numbers, and blood pressure. The investigators will compare improvements in heart disease risk factors and consumer satisfaction among the three HEP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Age 30-69 y;
* BMI: 25.0-37 kg/m2;
* Have hypercholesterolemia (total and LDL cholesterol 200-259 and 130-189 mg/dL, respectively),
* Systolic/diastolic blood pressure <140/90 mm Hg;
* Triglycerides <399 mg/dL, fasting glucose <109 mg/dL
* Body weight stable for 3 months prior (±3 kg);
* Stable physical activity regimen 3 months prior;
* Medication use stable for 6 months prior;
* Non-smoking;
* Non-diabetic;
* Not acutely ill;
* Females not pregnant or lactating;
* Participants must be willing and able to consume the prescribed diets and travel to testing facilities.

Exclusion Criteria:

* BMI <25 or >37
* Total cholesterol >259 mg/dL, low-density lipoprotein cholesterol >189 mg/dL,
* Triglycerides >400 mg/dL, fasting glucose >110 mg/dL
* Body weight changes in previous 3 months (±3 kg)
* Changes in physical activity regimen in the previous 3 months
* Medication changes in the previous 6 months
* Smoking
* Diabetic
* Acute illness
* Pregnant or lactating

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Risk factors for cardiovascular disease | 5 weeks
  Lipoprotein Particle Plus (LPP+) Panel. This comprehensive lipid panel will provide us with lipoprotein fractionation and particle number (VLDL, non-HDL, remnant lipoprotein, small/dense LDL III and IV, total measured HDL and LDL, and large buoyant HDL 2b), homocysteine, insulin, apolipoprotein A1, total apolipoprotein B, lipoprotein a, high sensitivity C-reactive protein, and a traditional lipid panel (total cholesterol, HDL cholesterol, calculated LDL cholesterol, triglycerides)

SECONDARY OUTCOMES:
Change in consumer perception and satisfaction of the HEPs | 5 weeks
  Consumer satisfaction and acceptance questionnaire. At the end of each dietary intervention, we will assess participants' satisfaction and acceptance of each HEP via an exit interview-style questionnaire
Risk factors for cardiometabolic disease | 5 weeks
  comprehensive metabolic panel which will include glucose, blood urea nitrogen (as a crude marker of protein intake), and markers of kidney and liver functions. Additionally, predictions of long-term cardiovascular disease risk and vascular age will be calculated using the Framingham Heart Study 10-year cardiovascular disease risk lipid equation.
Risk factors for cardiovascular disease | 5 weeks
  Change in diastolic and systolic blood pressure
Body weight | Measures will be taken twice per week throughout the entire enrollment period (15 weeks)
  Measures of weight in kilograms (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Campbell, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States